CLINICAL TRIAL: NCT06558227
Title: A Multicenter, Randomized, Open-label Phase II Study of ZG005 Combined With Bevacizumab Versus Sintilimab Combined With Bevacizumab for First-line Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Study of ZG005 Combined With Bevacizumab Versus Sintilimab Combined With Bevacizumab in Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-005
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Injections; Bevacizumab; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): ZG005 10 mg/kg administered intravenously every 3 weeks (Q3w) + Bevacizumab (Avastin®) 15 mg/kg administered intravenously Q3w
  Interventions: Biological: ZG005 for Injection; Biological: Bevacizumab
- Group B (Experimental): ZG005 20 mg/kg administered intravenously Q3w + Bevacizumab (Avastin®) 15 mg/kg administered intravenously Q3w
  Interventions: Biological: ZG005 for Injection; Biological: Bevacizumab
- Group C (Experimental): Sintilimab 200 mg administered intravenously Q3w + Bevacizumab (达攸同®) 15 mg/kg administered intravenously Q3w
  Interventions: Biological: Sintilimab; Biological: Bevacizumab

INTERVENTIONS:
Biological: ZG005 for Injection — 10 mg/kg or 20 mg/kg administered intravenously Q3w
  Other Names: ZG005
  Arms: Group A; Group B
Biological: Bevacizumab — 15 mg/kg administered intravenously Q3w
  Other Names: Avastin
  Arms: Group A; Group B
Biological: Sintilimab — 200 mg administered intravenously Q3w
  Arms: Group C
Biological: Bevacizumab — 15 mg/kg administered intravenously Q3w
  Other Names: 达攸同
  Arms: Group C

SUMMARY:
This study is a randomized, open-label, positive-controlled, multicenter phase II clinical trial. It evaluates the efficacy and safety of ZG005 combined with Bevacizumab compared to Sintilimab combined with Bevacizumab in first-line treatment for patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* 18-75 years of age;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1；
* Life expectancy ≥ 12 weeks.

Exclusion Criteria:

* Patients were deemed unsuitable for participating in the study by the investigator for any reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
progression free survival，PFS | through study completion, up to 2 year
  defined as the time from receiving treatment until disease progression or death from any cause, whichever happens first.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China